CLINICAL TRIAL: NCT03998995
Title: Virtual Reality Distraction From Procedural Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: J767 VR Children's Rehab; SCH2178 (Other: Sheffield Children's Hospital)
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Exostosis of Elbow; Upper Extremity Fracture; Burn; Arm; Burn Scald
Keywords: Immersive Virtual Reality (IVR); Patient-Centred Design; Upper Limb Injury; Children Rehabilitation
MeSH Terms: conditions — Burns; Arm Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVR rehabilitation game intervention (Experimental): Clinical trial patients' use the IVR rehabilitation game for two 15 minute sessions during one physical therapy session with their usual practitioner, with support from the physiotherapist and the game expert on the team.
  Interventions: Device: Immersive Virtual Reality

INTERVENTIONS:
Device: Immersive Virtual Reality — An Oculus Rift VR Headset and a set of Oculus Touch Controllers was used as interactivity device. Two scenarios of IVR rehabilitation game were offered to the patients: 1) Archery based on behind-the-neck overhead press, using a quiver on the user back to encourage bending their arm and firing the arrow to help with stretching exercises and 2) Climbing based on an overhead arm raise exercise.
  Each child will took part in a single IVR trial during their rehabilitation care with the physiotherapist, supported by IP, the games expert/researcher. Timing of participation was approximately 15 minutes of trial with each scenario of game. A short interview was conducted with each child and their parent (together) after each trial, and a focus group was conducted with the clinical staff.

SUMMARY:
This study explored the feasibility, acceptability and perceived the effectiveness of an Immersive Virtual Reality (IVR) 'game' in the rehabilitation of children with upper limb injuries. The objectives of the clinical trial were:

* To qualitatively assess the perceptions of child and parent regarding the acceptability of the game and equipment, and their perceptions of its effectiveness in reducing pain and discomfort and facilitating movement, compared to usual physical therapy experiences.
* To qualitatively assess physical therapy practitioners' perceptions of the effectiveness, usability, feasibility, and acceptability of VR in their clinical setting with this client group.

Hypothesis:

1. IVR rehabilitation game as an intervention will be acceptable to child patients and their parents.
2. IVR rehabilitation game experience will show less procedural pain, discomfort, and difficulties to movement, compared to usual physical therapy experiences.
3. IVR rehabilitation game will demonstrate any perceived disadvantages as a therapeutic intervention, compared with usual rehabilitation care.
4. IVR rehabilitation game will demonstrate usability in the clinical setting during the rehabilitation of a small sample of children with varying ULIs.

DETAILED DESCRIPTION:
Children with upper limb and hand injuries often have to undergo repetitive therapeutic exercises to regain or maximise function and movement which can be painful, uncomfortable and tedious, reducing compliance and limiting the movement and function achieved. There is a growing body of literature demonstrating the effectiveness of VR in reducing pain (e.g. in burns). Its effectiveness in rehabilitation, especially in children, is a promising but under-researched area. This study was focus on an under-researched target group in relation to IVR interventions, children undergoing physical therapies to enhance or optimise the upper limb and hand movement.

PARTICIPANT RECRUITMENT AND INFORMED CONSENT 10 children were recruited, plus one parent from each, and members of the clinical team of physiotherapists involved in their care. If considered suitable for the research, participants were introduced to the study and recruited via clinical staff responsible for their care. Staff was asked to provide information sheets to those who show interest in participation, including separate sheets for both child and parent.

If, having discussed the study with their child and other family members, parents were happy for their child to participate, and the child also wishes to participate, parents were asked to let a member of their clinical team know and arrangements were made for the date and time when the research will be take place.

Focus group: clinical staff involved in physical therapy for children where the VR intervention has been trialed was invited verbally, by letter or email to participate in a focus group after the trial is complete, and provided with an information sheet.

Having expressed an interest in hearing more about the study, based on a simple verbal explanation provided by staff, potential parents and children were provided with full, printed information (age-appropriate for children) about the study to read and consider in their own time. The information included a statement that participation is not obligatory and reassurance that refusal to participate will not affect their care, also explain that having decided to participate, the parent and child will be free to change their mind before, during or immediately after the study (prior to data analysis), without giving a reason. Advice was provided regarding how to withdraw their consent. Details regarding confidentiality, anonymity, data access, storage, and retention also were provided. It was suggested that the person retain the Information sheet for future reference and in order to make contact with the research team. Parents/children who, having read the information sheet and discussed the study together, wish to participate was asked to let the clinical staff know. Clinical staff contacted IP and made arrangements for him to visit the Unit on one of the child's appointment dates, to conduct the research. Shortly prior to using the VR for the trial on the day and before written consent was taken, the child was offered a 5-10 minute exposure to activities in the VR game (e.g. archery activity, rock climbing activity), to familiarise themselves, check there are no problems, and avoid unnecessary distractions and confusion during the procedure itself. If there were any problems or the child becomes unhappy about participation at this stage, they were reassured that they don't have to participate if they prefer not to and can also withdraw at any point during trial themselves if they wish. They were reminded verbally at this stage that deciding the study is not for them would have no consequences whatever for their future treatment.

If the child and their parent, having read the Information Sheet, expressed a wish to participate, tried out the equipment, and asked any questions they have, wish to go ahead, the parent was asked to sign a consent form and the child was asked to complete an assent form. This was done in the presence of a clinician on the research team, ahead of the intervention being implemented. Copies was be retained by the team, given to participants, with one copy kept in the child's medical notes.

DATA COLLECTION AND ANALYSIS A short interview was conducted with each child and their parent (together) after each trial and was audio recorded. These interviews took place in a quiet, private location near to where the physiotherapy and trial have taken place.

Focus groups with staff took place after all children's trials, in a quiet and private environment and at a time convenient for participants. Interviews and focus groups were guided by pre-written schedules and audio-recorded.

Thematic analysis was applied to all the resulting qualitative data, resulting from interviews with each child and parent, and focus group with therapeutic staff. This involved a process of careful reading, coding and comparison in order to identify important patterns in the data, focused on answering the aims of the study. Themes were generated based upon the analysis process, which were discussed and refined within the research team.

DATA HANDLING AND RECORD KEEPING On consenting to participate, participants were given a code (e.g. 01C, 01P for child01, parent01), by which they were identified for the duration of the study and in reports. A file linking participant identity to codes was created, password, and stored securely within a study file on a SHU password protected computer, as well consent forms. The lead investigator, IP, collect all data. He was audio record interviews and the focus group. Password protected digital recorders was used during interviews/focus groups to ensure data safety whilst on the ward and in transit back to the office. Recordings were saved as audio files on University-based password protected computers, then deleted. Audio files were used to create transcripts in the form of word documents, and both were securely stored in password protected computer files held by research team members. No one from outside the research team will have access to any information by which participant identity and data can be linked. The SHU and MRC Guidelines for research with human participants were followed in all aspects of the research, including data confidentiality. No one from the research team (who is not also a member of participants' clinical team) will require access to participants' medical records. Clinicians in the research team may make use of medical records - and their knowledge of their patients - in deciding whether to introduce the parent/child to the research study.

Consent forms are kept in locked cabinets in the locked office of the SHU-based project manager, SL. The cabinets themselves are kept locked (by key) at all times and only the key-holder will be able to access office and cupboards. Data collected for the study will be treated with the utmost care, retained within the research team, password protected/encrypted, and no one outside the team will have access. Personal information is securely stored within the SHU-based password protected computer files and separately from anonymised raw data. Files are password protected and encrypted for transfer.

Anonymised transcriptions made from the audio files and these are also saved as password protected files, identified by participant code. In reports, quotes from individuals will be only identified by participant code.

Throughout, data are stored securely and a study file maintained by SL. If the team is disbanded prior to this time, data will be stored at Sheffield Hallam University's research archive, SHURDA. Data will be collected and retained in accordance with the Data Protection Act 1998. All source documents will be retained for a period of 10 years following the end of the trial.

SAFETY ASSESSMENTS The Oculus Rift Virtual Reality headset was used with a laptop computer and all equipment was safety tested by the university before it used on participants. Appropriate health and safety measures were taken throughout the sessions, with each session limited to 15 minutes, with breaks in-between. Playing virtual reality games can sometimes cause disorientation, dizziness or nausea in some people, for example, those with severe motion sickness. However, in the most recent versions of this technology, and in our own recent trials of similar games, adverse reactions have been rare. Virtual rock climbing can also create anxiety in some children, especially if they suffer from vertigo. To check they were happy with the experience of VR before their sessions start, children were provided with a short 'test' session in the headset before parent and child agree to continue. Once the trial is underway, we asked the participating children to let us know straight away if they begin to feel uncomfortable or unwell.

The study was monitored and audited in accordance with the Monitoring Standard Operating Procedures of the Directorate of Research & Innovation at Sheffield Children's NHS Foundation Trust. All study related documents will be made available on request for monitoring and audits by the Sponsor, the Health Research Authority and the relevant Research Ethics Committee.

ETHICAL CONSIDERATIONS The study has been reviewed and approved by Sheffield Hallam University Research Ethics Committee, NHS Research Ethics Committee, and the Research and Development Dept. at Sheffield Children's Hospitals. The study was conducted in compliance with a Research Ethics Committee favourable opinion, Health Research Authority approval and Confirmation of Capacity & Capability at all participating sites.

The study was conducted in accordance with the International Conference for Harmonisation of Good Clinical Practice (ICH GCP), and the Research Governance Framework for Health and Social Care (2nd Edition).

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-16
* Upper limb or hand injuries, for which they are receiving rehabilitative care
* Able to speak and understand English

Exclusion Criteria:

* Injuries to the face or head that could hinder the correct positioning of the headset or pose an infection risk
* A learning impairment that could hinder the understanding of the task
* A history of severe motion sickness or vertigo.
* Mental health problems, such as anxiety.

Eligibility for parents:

* Having a child taking part in the study
* Being available on the day of treatment for interview
* Able to speak and understand English.

Eligibility for staff:

* Having a patient trialing VR during physiotherapy during which they were present as practitioner
* Being able to speak and understand English
* Being available on the day of the focus group

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Semi-structured interview with patients an family members | 10 minutes
  The interviews try to reflect on their experience using IVR concerning technology acceptance, emotional affect, usability and future deployment. In particular the interviews focused on four main areas: (1) the attitudes towards the VR rehabilitation session (e.g., "What did you like/dislike about the VR session compared to the normal therapy session?"); (2) the perceived difficulty and pain levels (e.g., "Compared to normal therapy sessions what was the pain you felt?"); the system usability / acceptability (e.g., "What is your overall impression regarding the VR rehabilitation?"); and the future VR deployment (e.g., "In the future, could you see this kind of therapy as a form of rehabilitation?").
Focus group with staff | 45 minutes
  The interviews try to reflect on their experience using IVR concerning technology acceptance, emotional affect, usability and future deployment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Children's Hospital, Sheffield, South Yorkshire, England, United Kingdom

REFERENCES:
- [Derived] Phelan I, Furness PJ, Matsangidou M, Carrion-Plaza A, Dunn H, Dimitri P, Lindley SA. Playing your pain away: designing a virtual reality physical therapy for children with upper limb motor impairment. Virtual Real. 2023;27(1):173-185. doi: 10.1007/s10055-021-00522-5. Epub 2021 Jun 9. PMID 36915630
- See also: IVR Children's Rehabilitation study: A presentation in the BBC Click program. — http://youtu.be/sDc5lIj1VbY?t=726